CLINICAL TRIAL: NCT05922488
Title: Effect of Umbilical Cord Milking Versus Delayed Clamping in Preterm Infants on Cerebral Oxygenation and Ductus Arteriosus Closure
Brief Title: Effect of Umbilical Cord Milking Versus Clamping in Preterms on Cerebral Oxygenation and Ductus Arteriosus Closure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, walaa M Madkoor, MD [walaa madkoor], Assistant fellow of pediatrics at Ahmed Maher teaching hospital, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: M D 75 / 2021
Record Dates: First submitted 2023-04-26; First posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Ductus Arteriosus
Keywords: Cerebral tissue oxygenation; Functional Ductus arteriosus closure; Umbilical cord milking; Delayed cord clamping
MeSH Terms: conditions — Ductus Arteriosus, Patent | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Intervention Model Description: all involved neonates will be randomized to DCC or UCM according to the randomization table and double-blinded method.
Masking Description: all involved neonates will be randomized to DCC or UCM according to the randomization table and double-blinded method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Umbilical cord milking (Experimental): In the cesarean section or vaginal delivery, the obstetrician will gently grasp the uncut umbilical cord and squeeze it from the placenta several times toward the infant usually within 20 seconds.
  Interventions: Procedure: Umbilical cord milking
- delayed cord clamping (Experimental): In the cesarean section or vaginal delivery the delivering obstetrician will wait at least 60 s before clamping the umbilical cord. Infants will be dried and will be given gentle tactile stimulation to promote the respiratory effort.
  Interventions: Procedure: delayed cord clamping

INTERVENTIONS:
Procedure: Umbilical cord milking — Umbilical cord milking : uncut umbilical cord and squeeze it from the placenta several times toward the infant usually within 20 seconds.
  Arms: Umbilical cord milking
Procedure: delayed cord clamping — delayed cord clamping: delivery the delivering obstetrician will wait at least 60 s before clamping the umbilical cord
  Arms: delayed cord clamping

SUMMARY:
All patients will be subjected to the following:

1-Umbilical cord milking or delayed cord clamping according to the ranamization table 2 serial measurement of cerebral tissue oxygenation 3- serial echocardiography for ductus arteriosus (DA)functional closure

DETAILED DESCRIPTION:
* Study Population: neonates born and admitted to Ain shams university neonatal intensive care units (NICUs).

  * Inclusion criteria:

    o Preterm infants with gestational age (GA) of 28 - 34 weeks born and admitted to Ain shams university NICUs.
  * Exclusion criteria:

    * Late preterm with gestational age 34-37 weeks.
    * Term infants with gestational age > 37 weeks.
    * NIRS data that was not obtained within 1st hour after birth.
    * Congenital heart disease (other than DA or small atrial septal defects/patent foramen oval/ventriculi septal defects).
    * Hypoxic-ischemic insult.
    * Major congenital deformations. #All participants will be subjected to the following:
* Infants will be considered to be randomized at the time of enrolment for:

  o Delayed cord clamping (DCC) and Umbilical cord milking (UCM)
* Near-infrared spectroscopy (NIRS):

  * In the delivery room: after the intervention (UCM or DCC) the regional cerebral tissue oxygenation (rScO2 ) and cerebral fractional tissue oxygen extraction (c FTOE) will be collected for 10 minutes within 1st hour after birth.
  * In the neonatal intensive care unit: NIRS data will be collected for 2 hours at 12,24 hours, and 48 hours after birth.
* Echocardiography:

will be performed at 6, 12, 18, 24, and 48 hours of life by using an ultrasound Doppler machine Mindary.M9. assessment of DA functioning closure by measuring duct diameter and direction of blood flow through it.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants with gestational age (GA) of 28 - 34 weeks born and admitted to Ain shams university NICUs.

Exclusion Criteria:

* Late preterm with gestational age 35-37 weeks.

  * Term infants with gestational age > 37weeks.
  * NIRS data that not obtained within 1sthour after birth.
  * Congenital heart disease (other than PDA or small atrial septal defects/patent foramen oval/muscularventriculoseptal defects).
  * Hypoxic-ischemic insult.
  * Major congenital deformations.

Max Age: 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
time of functional ductus arteriosus closure | 6, 12, 18, 24, and 48 hours of life
  performed by follow-up echocardiography using machine Mindary.M9 measuring changes from the baseline blood flow direction through the ductus arteriosus (DA) at 6, 12, 18, 24, 48 hours of life that helps to determine at which time the functional closure of ductus arteriosus occurs.

SECONDARY OUTCOMES:
changes in cerebral tissue oxygenation by NIRS. | First hour of life for 10 minutes/ and for 2 hours on 12,24,84 hours of life
  Cerebral tissue oxygenation measurement using Near-infrared spectroscopy (NIRS):
  * In the delivery room: after the intervention (UCM or DCC), rScO2 and cFTOE will be collected for 10 minutes within 1st hour after birth.
  * In the neonatal intensive care unit: NIRS data will be collected for 2 hours at 12,24 hours, and 48 hours after birth.
ductus arteriosus diameter | 6, 12, 18, 24, and 48 hours of life
  performed by follow-up echocardiography at 6, 12, 18, 24, and 48 hours of life by using an ultrasound Doppler machine Mindary.M9 comparing changes that occur in the ductus arteriosus diameter from the baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Ainshams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No